CLINICAL TRIAL: NCT06754696
Title: Evaluation of Blood Protein O-GlcNAcylation Levels in Children - CHANCE Study (Child Heart O-glcnAc Nantes)
Brief Title: Evaluation of Blood Protein O-GlcNAcylation Levels in Children
Acronym: CHANCE
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0573
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Septic Shock; Development and Health; Metabolism Changes
Keywords: O-GlcNAcylation; Sepsis; Septic shock; metabolism; children
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy group: children attending hospital and receiving a blood sample as part of their care during general paediatric consultations, anaesthesia or day hospital consultations.
  Children requiring a blood test as part of a medical indication in the first week of life / blood samples taken at birth from cord blood.
  A blood sample will be taken at inclusion during a blood test carried out in the care unit, and possibly if other blood samples are planned as part of the care, additional samples will be taken in a maximum of 6 tubes in 48 hours, i.e. for a total volume of 600 µl to 3 ml. The child's clinical data will be collected in his medical file.
- Septic shock: Children attending a paediatric emergency department for a severe infection requiring vascular filling, or a child admitted to an intensive care unit for sepsis or presenting with sepsis during hospitalisation.
  A blood sample will be taken at inclusion during a blood test carried out in the care unit and then at H3, H6, H12, H24 and H48, i.e. 6 times in 48 hours for a total volume of 600 µl to 3 ml for patients in septic shock. The child's clinical data will be collected in his medical file.

SUMMARY:
Stimulation of O-GlcNAcylation has been shown to be beneficial in several acute pathologies and different animal models, such as haemorrhagic and septic shock, and ischaemia-reperfusion (cerebral and cardiac). It could therefore be interesting to use this approach in children in order to limit the impact of various pathologies inducing SIRS, such as extracorporeal circulation for major surgery, septic shock or various traumas. The investigators demonstrated in 2 different animal models (endotoxemia by injection of Lipopolysaccharides and caecal puncture ligation model) with 3 different pharmacological molecules (Glucosamine, ThiametG and NButGT) that stimulation of O-GlcNAcylation was beneficial in the early phase of septic shock with a marked effect on cardiac function and survival. The investigators thus demonstrated that stimulation of O-GlcNAcylation was beneficial in young rats in septic shock. However, none of this work has yet been reproduced in humans, either children or adults.

DETAILED DESCRIPTION:
Sepsis is a major but potentially preventable cause of death in children worldwide, with a mortality rate of 29%. It also causes 28% of mild disability and 17% of severe disability in Europe. It is important to note that most studies only look at septic shock in adults, but the populations most affected by septic shock are young children and the elderly. An obvious difficulty in the diagnosis of septic shock in paediatrics is related to the variability of physiological values according to age and the specific pathophysiological features of this pathology in children. Septic shock should be suspected when the child presents with a change in mental status associated with infection and signs of tissue hypoperfusion. Unlike in adults, where septic shock is classically biphasic with an early phase of vasoplegia followed by a phase of low cardiac output, a specific haemodynamic profile is observed in children. It is characterised by severe hypovolemia requiring vascular filling with very heterogeneous responses, low cardiac output and high systemic arterial resistance. In children, septic shock is a dynamic process with heterogeneous haemodynamic phases that change during the course of the shock. The therapeutic agents used and their doses must therefore be adjusted at all times to maintain vascular perfusion. Between 2005 and 2011, more than half of paediatric deaths from septic shock occurred within the first 24 hours. Prompt treatment is a vital factor in the prognosis, with each additional hour spent in shock doubling the risk of death. Unlike in adults, low cardiac output, rather than increased systemic vascular resistance, is associated with mortality. Due to a higher basal heart rate, the increase in heart rate is more limited than in adults. Although the physiopathology of children is different (lower cardiac reserve, lower basal arterial pressure), there are no specific recommendations for children; those for adults are adapted to this population. On the basis of these alarming data, there is a significant socio-economic interest in identifying new treatments for the management of young patients.

Cardiac metabolism is an important area of research because it plays a central role in maintaining cardiac function under stress. In recent years, O-N-acetyl-glucosaminylation, more simply known as O-GlcNAcylation, a post-translational modification of proteins, has attracted considerable interest because it plays a key role in regulating cellular metabolism, but also in the ability to adapt to stress and cell survival. Particular attention has been paid to this metabolic pathway in various pathologies (Alzheimer's disease - patent US20200079766, diabetes, heart attack, etc.) but always in adults or the elderly. The work that investigators have carried out shows that the levels of O-GlcNAcylation of cardiac proteins vary during the early stages of life in rats. This observation is crucial because it could explain some of the metabolic peculiarities of the young heart (use of mainly glycolytic substrates during the first days of life, for example) and the greater capacity of the hearts of newborn rats to withstand stress such as ischaemia-reperfusion. O-GlcNAcylation is a ubiquitous, rapid and reversible post-translational modification involving the addition of a monosaccharide: ß-D-N-acetylglucosamine to the serine and threonine residues of proteins. In physiological conditions, 2 to 3% of the glucose entering the cell is directed towards the hexosamine biosynthesis pathway (VBH), which leads to the production of UDP-GlcNAc used by O-GlcNAc transferase (OGT) to O-GlcNAcylate proteins. The reverse reaction is catalysed by O-GlcNAcase (OGA). VBH is at the crossroads of several cellular metabolic pathways (glucose, acetyl-CoA, glutamine, uridine and ATP) and O-GlcNAcylation is considered to be a metabolic sensor. The number of O-GlcNAcylated targets (+8000 proteins) bears witness to the involvement of this modification in various cellular functions. O-GlcNAc levels are finely modulated according to the cell's metabolic environment, enabling it to adapt to stress. This last point is particularly important as metabolism changes during development, and could have an impact on the hexosamine biosynthesis pathway and therefore on O-GlcNAcylation. Stimulation of O-GlcNAcylation has been shown to be beneficial in several acute pathologies and different animal models. It could therefore be interesting to use this approach in children to limit the impact of various pathologies that induce SIRS, such as extracorporeal circulation for major surgery, septic shock and various traumas.

ELIGIBILITY:
1. Healthy group

   Inclusion Criteria :
   * Age from 0 to 17 years at the time of sampling (including premature infants)
   * Children coming to hospital for a blood sample to be taken as part of a pre-operative check-up, an allergy check-up or a check-up as part of a pathology other than sepsis.
   * Premature infants benefiting from a blood sample as part of their monitoring and management of prematurity
   * Collection of umbilical cord blood
   * Signed consent

   Exclusion Criteria :
   * Children with an infection
   * Children with fever
   * Children with an immune deficiency
   * Children with autoimmune disease
   * Children with metabolic disease
   * Children with haematological diseases
   * Children with a genetic disease
   * Unsigned consent
   * Refusal by parents or child
2. Septic group

Inclusion Criteria :

* Age from 0 to 17 years at the time of sampling (including preterm infants)
* Children with suspected sepsis or diagnosed sepsis according to the 2016 definition
* Premature infants having blood drawn for suspected or diagnosed sepsis
* All responsible bacteria, viruses or fungi
* Signed bio-collection consent

Exclusion Criteria :

* Children with an immune deficiency
* Children with autoimmune disease
* Children with a metabolic disease
* Children with haematological diseases
* Children with a genetic disease
* Unsigned bio-collection consent
* Refusal by parents or child

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All children attending hospital and receiving a blood sample as part of their care during general paediatric consultations, anaesthesia or day hospital consultations.
  Children attending a paediatric emergency department for a severe infection requiring vascular filling, or a child admitted to an intensive care unit for sepsis or presenting with sepsis during hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2036-01-31 (Estimated); Study Completion 2036-01-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of O-GlcNAcylation levels in children | At inclusion
  Assess protein O-GlcNAcylation levels as function of age
Assess the impact of septic shock on O-GlcNAcylation levels: - Comparison of O-GlcNAcylation levels between healthy patients and patients in septic shock | Between inclusion and 48 hours after inclusion
  Comparison of O-GlcNAcylation levels between healthy patients and patients in septic shock

SECONDARY OUTCOMES:
Analysis of a potential link between O-GlcNAcylation levels and the prognosis of patients in septic shock | Up to 5 years after inclusion
  Study of the correlation between O-GlcNAcylation levels and the prognosis of patients in septic shock

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided